CLINICAL TRIAL: NCT05847231
Title: The Effect of Mandala Coloring Applied to Caregivers Caring for Palliative Care Patients on Perceived Stress, Anxiety Level, and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/ 05- 08
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Perceived Stress; Anxiety Level; Quality of Life
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Intervention Model Description: Mandala
Who Masked: Participant
Masking Description: Single (Participant) Perceived Stress, Anxiety Level and Quality of Life
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mandala app (Experimental): mandala will be aplicated
  Interventions: Behavioral: Perceived Stress, Mandala application
- routine maintenance practice (No Intervention): Routine maintenance will be applied.

INTERVENTIONS:
Behavioral: Perceived Stress, Mandala application — Mandala
  Other Names: Anxiety Level; Quality of Life
  Arms: mandala app

SUMMARY:
The word palliative comes from the Latin word "pallium" meaning "cover". The aim of palliative care is not to eliminate the cause of the disease; to alleviate the negative effects of the disease.

Mandala painting, which is one of the non-pharmacological applications, is an art therapy technique that can provide psychological support and healing. Mandala painting is a safe and accessible activity that requires no special skills and can be used as a complementary strategy to support mental health. In the literature, it is stated that coloring mandala improves psychological symptoms and relieves the person. The artistic view of nursing is to understand the needs of the individual, the sources of anxiety, anxiety and stress, and then to develop practices that will increase his/her self-confidence and resilience by increasing his/her ability and competence level. Therefore, this study was planned to examine the effect of mandala painting applied to caregivers caring for palliative care patients on perceived stress, anxiety level and quality of life.

This research, which is planned as a randomized experimental study with pretest-posttest control group, will be a study for informal caregivers who have patients in the palliative service of fethi sekin city hospital between May 2023 and December 2023. The sample will consist of 80 (40 experimental, 40 control) caregivers who accepted the research that met the research criteria.

Experimental group will be composed of caregivers who will paint mandalas. In addition to verbal and written information, the Patient Description Form, Perceived Stress Scale (PSÖ), State-Trait Anxiety Scale (WHO) and Short Form (SF-36) Quality of Life Scale have been applied to the 1st Stage. measurement will be obtained. The program will be implemented for 4 weeks, 4 days a week. 16 pre-selected mandala drawings will be printed separately on A4 papers and a new drawing will be given to caregivers every week. Mandala coloring papers and 12 colored felt-tip crayons will be given to each participant by the researcher. After the end of the sessions, the second measurements will be obtained by applying the Perceived Stress Scale (PSS), State-Trait Anxiety Scale (DSQ) and Short Form-36 (SF-36) Quality of Life Scale.

DETAILED DESCRIPTION:
The palliative care approach first emerged in the 11th century as a religious-based volunteer movement for the treatment of people suffering from terminal illnesses during long journeys. Although the quality of patient care changes all over the world, there is definitely a section in care that includes the responsibilities of the family. It is stated in the literature that the anxiety levels of the patient and family members who receive the necessary information and support about the disease decrease. The caregiving process is a very stressful situation for the caregiver, which can lead to physical and psychological problems. Anxiety levels of caregivers also increase due to the caregiving process that creates excessive stress and anxiety. Studies in which caregivers have high levels of anxiety due to the burden of care come to the fore in the literature. Mandala provides calming and relaxation as your mind. It silences the negative and complex emotions that bother the person himself. With the relaxation it provides, it allows the individual to listen to himself and to rest spiritually. Mandala allows to see holistically. While increasing one's awareness, it reveals what is hidden in the unconscious. Art therapy helps individuals feel themselves at the center of their lives, express themselves and discover who they are in the group while drawing, painting or making mandalas.

Jung stated that he created mandalas in times of distress when both he and his patients felt negative emotions. İn the previous studies; Mandala art therapy has been used to define psychiatric problems in children, to reduce stress and to calm down, to provide concentration and psychological relaxation, and positive results have been obtained.

ELIGIBILITY:
Inclusion Criteria:

* be over 18 years old
* Palliative care patient being the only informal caregiver
* There is no physical problem that will prevent painting mandala. (seeing, hearing, etc.)
* Being able to use their hands actively
* No communication problem
* No learning problems
* Being suitable/willing to work with the group

Exclusion Criteria:

* be under the age of 18
* Palliative care patient is not the only informal caregiver
* Having a physical problem that will prevent you from painting a mandala (sight, hearing, etc.)
* Having a physical disability in the upper extremity of the caregiver
* Having trouble communicating
* Having a learning problem
* It does not show the harmony of working with the group.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS)Perceived Stress Scale (PSS) | after 1 hour in mandala app
  It is designed to measure how stressful individuals perceive their experiences, including their feelings and thoughts that they may have experienced during the last month. The total score that can be obtained from the scale is 32. The scale consists of 8 items. These items are scored by the individual in a 5-point Likert type (0=Never,1=Rarely,2=Sometimes,3=Frequently, 4=Very often) according to their intensity of experience. While five items of the scale are plain (1st, 2nd, 3rd, 7th, 8th items); three items are reversed (items 4, 5, 6). It has two subscales: perceived stress (1st, 2nd, 3rd, 7th, 8th items) and perceived coping (4th, 5th, 6th items).

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (WHO) | after 1 hour in mandala app
  n this study, the part of the scale measuring trait anxiety was used to determine the trait anxiety levels of the patients. Trait Anxiety Inventory is a 4-point Likert-type with 20 items and is scored as "never": 1, "a little": 2, "a lot": 3, "completely": 4, according to the degree of severity of the feelings, thoughts or behaviors expressed by the items. . There are direct or reverse scored statements in the scale. Reverse scored statements; Items 1, 6, 7, 10, 13, 16 and 19. Trait anxiety score is obtained by adding the constant value of 35, which is the constant value of the trait anxiety scale, to the value obtained by subtracting the total score of the reverse scored statements from the total score of the direct statements. The lowest score that can be obtained from the scale is 20, and the highest score is 80. A high score indicates a high level of anxiety, a low score indicates a low level of anxiety.

OTHER OUTCOMES:
SF-36 Quality of Life Scale | after 1 hour in mandala app
  The scale consists of 36 questions and consists of physical functionality (10 questions), social functionality (2 questions), physical role restrictions (4 questions), emotional role restrictions (3 questions), mental health (5 questions), energy/vitality (4 questions), pain (2 questions), general health perception (5 questions). The answers to the questions are in 2, 3, 5, and 6 point likert type. Scoring of the scale takes place in two stages. In the first stage, 0 represents the lowest quality of life value and 100 represents the highest quality of life value. In the second stage, scores for each dimension are obtained. A score close to 0 indicates undesirable poor health, and closer to 100 indicates desired good health.

CONTACTS AND LOCATIONS:
Locations (1):
- Gülcan B.Turan, Elâzığ, Merkez, Turkey (Türkiye)